CLINICAL TRIAL: NCT06841874
Title: Expanded Access Program of Taletrectinib in Patients With Advanced or Metastatic ROS1-Positive NSCLC
Acronym: Tale EAP
Status: No longer available | Type: Expanded Access
Sponsor: Nuvation Bio Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AB-106-EAP
Record Dates: First submitted 2025-02-11; First posted 2025-02-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Carcinoma; Bronchogenic Carcinoma; Non Small Cell Carcinoma of the Lung; ROS1-positive Non-Small Cell Lung Cancer (NSCLC)
Keywords: Non-Small Cell Lung Cancer (NSCLC); ROS1-Positive Non-Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Carcinoma; Carcinoma, Bronchogenic; Carcinoma, Non-Small-Cell Lung | interventions — taletrectinib

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Taletrectinib — Oral capsule
  Other Names: AB-106

SUMMARY:
This Expanded Access Program will provide access of taletrectinib therapy to patients with locally advanced or metastatic ROS1-positive NSCLC who are not an appropriate candidate for an approved therapy, for any ongoing taletrectinib clinical trial and who, in the opinion of their oncologist, may benefit from treatment.

DETAILED DESCRIPTION:
This Expanded Access Program will provide access of taletrectinib therapy to patients with locally advanced or metastatic c-ros-oncogene 1 (ROS1)-positive non-small cell lung cancer (NSCLC). These patients are not an appropriate candidate for an approved therapy, including crizotinib, entrectinib, or repotrectinib, for participating in ongoing Nuvation Bio clinical trial AB-106-G208 and who, in the opinion of their oncologist, may benefit from treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically or cytologically confirmed diagnosis of locally advanced (including inoperable Stage IIIA or IIIB NSCLC) or metastatic NSCLC.
* Evidence of ROS1 gene fusion.
* Adequate bone marrow and organ function
* Ineligible for participation in ongoing Nuvation Bio clinical trial AB-106-G208. Exception may be granted by the Sponsor/Supplier if they have a restriction or hardships that prevent them from participating in a clinical trial.
* Failed approved therapy or are not an appropriate candidate for an approved therapy including crizotinib, entrectinib, or repotrectinib.

Exclusion Criteria:

* Prior systemic anticancer therapy washout of 5 half-lives or 2 weeks, whichever is sooner.
* Patients who develop acute medical conditions which require immediate treatment or stabilization (e.g., new diagnosis of pulmonary embolism that requires anti-coagulation; acute and symptomatic spinal cord compression that requires immediate spinal radiotherapy). Note: patients may enroll after starting treatment for these acute conditions and the patients are considered stabilized.
* History or evidence of interstitial fibrosis, interstitial lung disease or drug-induced pneumonitis that did not resolve prior to screening.
* Active and untreated hepatitis B or C. Exception is chronic stable hepatitis B and C with stable liver function at screening.
* Ongoing cardiac dysrhythmias of Common Terminology Criteria for Adverse Events (CTCAE) ≥Grade 2, uncontrolled atrial fibrillation of any grade, or QT interval corrected for heart rate by Fridericia's formula >470 milliseconds, or symptomatic bradycardia <45 beats per minute; patient has family or medical history of long QT syndrome.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult